CLINICAL TRIAL: NCT03294473
Title: Centralized IIS-Based Reminder Recall to Increase Influenza Vaccination Rates in New York State - Second Trial in New York State
Brief Title: Centralized Reminder Recall - Flu RCT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); New York State Department of Health (Other Government); University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Peter G Szilagyi, MD MPH, Executive Vice Chair, Clinical Research, UCLA David Geffen School of Medicine, Dept of Pediatrics, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 17-001153; 1R01AI114903 (NIH); 17-001153 (Other: University of California, Los Angeles, IRB)
Record Dates: First submitted 2017-09-22; First posted 2017-09-27 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Influenza, Human; Orthomyxoviridae Infections; RNA Virus Infections; Virus Disease; Respiratory Tract Infections; Respiratory Tract Disease; Vaccines; Physiological Effects of Drugs
Keywords: reminder recall (R/R), influenza vaccines
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections; RNA Virus Infections; Virus Diseases; Respiratory Tract Infections; Respiratory Tract Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Autodial R/R (Experimental): R/R Autodialers:Participants in this group will receive up to 3 influenza vaccination reminders via telephone call - with a brief educational message + practice name + practice phone number
  Interventions: Behavioral: R/R - Autodialers
- Text Message R/R (Experimental): R/R Texting: Participants in this group will receive up to 3 influenza vaccination reminders via text message - with a brief educational message + practice name + practice phone number
  Interventions: Behavioral: R/R - Texting
- Postcard R/R (Experimental): R/R Mailed Postcard:Participants in this group will receive up to 3 influenza vaccination reminders via postcard - with a brief educational message + practice name + practice phone number
  Interventions: Behavioral: R/R - mailed postcard
- Standard of Care Control (No Intervention): Participants in this group will not receive any influenza vaccination reminders

INTERVENTIONS:
Behavioral: R/R - Autodialers — Investigators will send out flu vaccine reminder recall notices via autodialer message to the parents of children 6 months - 17 years of age who are due for the flu vaccine, per the records in the New York State Immunization Information System (NYSIIS).
  Arms: Autodial R/R
Behavioral: R/R - Texting — Investigators will send out flu vaccine reminder recall notices via text message to the parents of children 6 months - 17 years of age who are due for the flu vaccine, per the records in the New York State Immunization Information System (NYSIIS).
  Arms: Text Message R/R
Behavioral: R/R - mailed postcard — Investigators will send out flu vaccine reminder recall notices via mailed postcards to the parents of children 6 months - 17 years of age who are due for the flu vaccine, per the records in the New York State Immunization Information System (NYSIIS).
  Arms: Postcard R/R

SUMMARY:
This study is related to a previous study, Clinicaltrials.gov ID: NCT02924467. There are some modifications in relation to the intervention arms as well as the use of a different cohort, thereby justifying the second submission to Clinicaltrials.gov. This trial is taking place in New York State, through partnership with the New York State Health Department (excluding New York City), and Colorado. Each state will have it's own Clinicaltrial.gov submission -- this was decided as some of the intervention components are different enough that separate registrations were warranted.

Despite U.S. guidelines for influenza vaccination of all children starting at 6 months, only about half of children are vaccinated annually leading to substantial influenza disease in children and spread of disease to adults. A major barrier is that families are not reminded about the need for their children to receive influenza vaccination. The investigators will evaluate the impact of patient reminder/recall (R/R) performed by state immunization information systems to improve influenza vaccination rates by using 4 clinical trials (2 per state) in two different states. The investigators will assess effectiveness and cost-effectiveness of 1) autodialer R/R 2) text messages R/R 3) mailed postcard R/R as compared to 4) standard of care control (no R/R).

DETAILED DESCRIPTION:
Annual epidemics of influenza A and B cause substantial morbidity and mortality in the US with high rates of hospitalizations, emergency department visits, outpatient visits, and medical costs. Epidemics cause up to 40,000 deaths/year (mostly elderly) and extensive morbidity among children who play a key role in instigating and expanding epidemics. In addition, concerns about pandemic influenza heighten the importance of new mechanisms to rapidly inform the population about influenza and direct efforts for rapid vaccine delivery.

Since 2010, the Advisory Committee on Immunization Practices (ACIP) has recommended influenza vaccination for all children >6 months of age. However, vaccination rates remain very low. For the 2012-2013 season, only 56% of children 2-17years were vaccinated. Modeling studies suggest that as many as 19 million cases of influenza could be prevented if child vaccination rates were raised to 70% nationally.

The most effective strategy recommended by CDC and the Task Force on Community Preventive Services for improving childhood influenza vaccination rates is reminder/recall (R/R), sent by phone or mail, notifying parents of the need to vaccinate their child. We and others have shown that R/R can improve influenza vaccination rates by up to 20%. However, <16% of practices use R/R; barriers are practice costs, insufficient staff time and expertise, and lack of predictability regarding receipt of vaccine supplies.

Statewide immunization information systems (IISs) now exist in all states to track childhood vaccinations, but they have not been used for influenza vaccine R/R because of lack of evidence for their effectiveness and a lack of a template for IIS-based R/R. The investigators have united two leading immunization research groups (Denver, CO and Rochester (lead by personnel at UCLA), NY) to assess the impact of centralized IIS-based influenza vaccine R/R and to evaluate the effect of three types of R/R (autodialer, text message and mail R/R) over usual care. The investigators will also develop tools to aid other states in creating efficient IIS R/R systems for seasonal and possible pandemic influenza outbreaks.

For this second R/R trial in New York State, the intent is to evaluate the impact of reminder recalls, in the form of 1) autodialers 2) text messages and 3) postcards versus the standard of care control group, specifically in relation to raising influenza vaccination rates among children 6m-17 years of age.

The proposed design of this 4-arm RCT:

1. standard of care control
2. autodialer R/R -- with brief educational messages, practice name and practice phone number
3. text message R/R-- with brief educational messages, practice name and practice phone number
4. mailed (postcards) R/R-- with brief educational messages, practice name and practice phone number

Hypothesis 1: All IIS-C R/R modalities will be more effective than usual care

Hypothesis 2: Text messaging will be more cost-effective than other modalities

ELIGIBILITY:
Inclusion Criteria:

* a record in the New York State Immunization Information System
* in need of at least one influenza vaccination at the time of the beginning of the study
* affiliated with a participating practice (145 randomly selected)

Exclusion Criteria:

* no record within the New York State Immunization Information System
* up to date on their influenza vaccination
* not affiliated with an eligible practice

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70190 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2018-04-19 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome is receipt of influenza vaccine comparing effectiveness of standard of care control to autodialer, text message and postcard R/R | 6 months
  Based on our prior studies, we plan to send up to 3 autodialer, text messages or postcards (based on randomization) reminders, roughly every 5-6 weeks. This will begin in October 2017 and end in December 2017. Outcomes are assessed at 6 months using IIS data.

SECONDARY OUTCOMES:
Cost of the R/R intervention | 6 months
  A cost-effectiveness analysis will be conducted to determine which modality of R/R (autodialer, text message or mailed postcard) is the most cost-effective in relation to improving influenza vaccination rates. The cost analysis will also compare autodialer to text, autodialer to postcard, and texting to postcards.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Szilagyi, MD, MPH, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate results will be prepared for publication at the end of the trial.

REFERENCES:
- [Derived] Szilagyi PG, Albertin CS, Saville AW, Valderrama R, Breck A, Helmkamp L, Zhou X, Vangala S, Dickinson LM, Tseng CH, Campbell JD, Whittington MD, Roth H, Rand CM, Humiston SG, Hoefer D, Kempe A. Effect of State Immunization Information System Based Reminder/Recall for Influenza Vaccinations: A Randomized Trial of Autodialer, Text, and Mailed Messages. J Pediatr. 2020 Jun;221:123-131.e4. doi: 10.1016/j.jpeds.2020.02.020. PMID 32446470